CLINICAL TRIAL: NCT01833819
Title: Opioid-free Total Intravenous Anesthesia With Propofol, Dexmedetomidine and Lidocaine Infusions for Laparoscopic Cholecystectomy; Comparison With Propofol, Remifentanil Infusions
Brief Title: Anesthesia With Propofol, Dexmedetomidine and Lidocaine Infusions for Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.BAV.0.05.05/346
Record Dates: First submitted 2013-03-12; First posted 2013-04-17 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Cholecystitis
Keywords: Laparoscopic cholecystectomy,; Total intravenous anesthesia,; Propofol,; Dexmedetomidine,; Lidocaine,; Remifentanil,; Postoperative analgesic consumption,; Postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Lidocaine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opiod-free group (Other): Opioid-free anesthesia (Group DL) with dexmedetomidine (0.6 mg/kg loading, 0.3 mg/kg/h infusion), lidocaine (1.5 mg/kg loading, 2 mg/kg/h infusion), and propofol infusions (3-12 mg/kg/h).
  Interventions: Drug: Dexmedetomidine and lidocaine
- Opioid-based group (Other): Opioid-based anesthesia (Group RF) with single dose fentanyl (2μg/kg), remifentanil (0.25μg/kg/min), and propofol infusions (3-12 mg/kg/h).
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine and lidocaine
  Arms: Opiod-free group
Drug: Remifentanil
  Arms: Opioid-based group

SUMMARY:
Opioids may attenuate postoperative hyperalgesia and postoperative nausea and vomiting. Our hypothesis is: opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy may achieve comparable hemodynamic stability during laparoscopy, with lower postoperative analgesic consumption and incidence of postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Patients are randomly allocated into two groups to have either opioid-free anesthesia (Group DL) with dexmedetomidine (0.6 mg/kg loading, 0.3 mg/kg/h infusion), lidocaine (1.5 mg/kg loading, 2 mg/kg/h infusion), and propofol infusions or opioid-based anesthesia (Group RF) with fentanyl, remifentanil (0.25μg/kg/min), and propofol infusions.

Simple randomization was done using 80 opaque sealed envelopes, 40 for each group, indicating group assignment and describing the anesthetic protocol. Before anesthesia induction, an anesthesiologist will open the next envelope in the sequence to reveal the treatment allocation. This anesthesiologist will only prepare the study medications and will be involved in neither preoperative and postoperative data collection nor anesthesia management of the patients.

The drugs will be delivered in 10 ml and 50 ml syringes labeled as "loading" or "infusion" respectively. To ensure proper blinding, the loading doses of drugs (dexmedetomidine and lidocaine in Group DL or fentanyl and normal saline in Group RF) will be calculated according to the patient's body weight and diluted to a 10 ml volume labeled as "loading-1" and "loading-2" in order of administration. The infusion drugs (dexmedetomidine and lidocaine in Group DL or remifentanil and normal saline in Group RF) will be prepared in 50 ml syringes and labeled as "infusion-1" and "infusion-2" respectively.

At the preoperative holding area, patients will be instructed in the use of the verbal numerical rating scale (VNRS) and patient controlled analgesia (PCA) pump. Same anesthesiologist (MB) who is blinded to the study groups will perform the anesthesia management of all procedures.

On arrival at the operating room, standard monitoring will be applied consisting of ECG, noninvasive blood pressure, pulse oximetry and bispectral index (BIS). After premedication with intravenous midazolam (0.03 mg/kg), baseline heart rate and mean arterial blood pressure (MAP) will be determined which are average of three consecutive measurements. Preoxygenation with 5 L/min of pure oxygen will be performed during administration of loading doses. Before induction, patients in Group DL received 0.6 μg/kg dexmedetomidine (loading-1) diluted to a total volume of 10 ml and infused in 10 minutes. To avoid bias, patients in Group RF will receive 2 μg/kg fentanyl in same fashion. At the induction, dexmedetomidine or remifentanil (1 μg/ml and 50 μg/ml respectively, infusion-1) infusions 0.3 ml/kg/h will be started and lidocaine 1.5 mg/kg (loading-2) in Group DL or normal saline in Group RF and propofol 1.5 mg/kg will be administered. Lidocaine (20 mg/ml) or normal saline infusions 0.1 ml/kg/h and propofol infusion 10 mg/kg/h will be started immediately after loading doses. Vecuronium 0.1 mg/kg i.v. will be given to facilitate tracheal intubation.

The lungs will be mechanically ventilated with a mixture of oxygen in air (FiO2: 50%, tidal volume 7-10 ml/kg, respiratory rate 10-14/min) to obtain an end-tidal CO2 (EtCO2) value between 30-35 mmHg. Supplemental neuromuscular blockade will be achieved with vecuronium after assessment of neuromuscular function with train-of-four.

Dexmedetomidine and lidocaine infusions in Group DL or remifentanil and normal saline infusions in Group RF will kept constant during surgery. Propofol infusion rate will be adjusted 3-12 mg/kg/h to maintain the MAP within ±20% of the baseline value, and to maintain a BIS reading below 50. The lidocaine or normal saline administration will be terminated after gallbladder extraction (or 10 min before the end of surgery). Dexmedetomidine or remifentanil and propofol administration will be terminated during skin closure.

All patients in both groups will receive 8 mg dexamethasone and 50 mg dexketoprofen trometamol i.v. after anesthesia induction and 1 g paracetamol i.v. after gallbladder extraction. Laparoscopic portals will be infiltrated with 20 ml 0.5% bupivacaine including 1/80.000 adrenaline before skin closure.

Surgery: Surgeons who are experienced in laparoscopic cholecystectomy will performed the operations using standard 4-trocar technique. A blunt-tipped 12-mm trocar will be used to access the peritoneal cavity. Pneumoperitoneum will be achieved with carbon dioxide, and intra-abdominal pressure will be maintained at 12-14 mmHg throughout surgery. Three additional 5-mm ports will be introduced and patients will be positioned in 30 degrees anti-Trendelenburg position and be rotated toward the left side to facilitate exposure of the gallbladder. After endotracheal intubation a nasogastric tube will be inserted and stomach content will be aspirated. At the end of surgery, the inflated carbon dioxide will carefully be evacuated by manuel compression of the abdomen.

A PCA pump will be ready to use immediately after extubation. The PCA pump will set to deliver fentanyl i.v. with a bolus dose of 20 μg, a lock-out of 5 min, without continuous infusion and dose limit for 6 hours after surgery. Trained nurses, blinded to treatment allocation and with no access to the intraoperative records, will perform all outcome assessments in the postanesthesia care unit (PACU) and surgical ward. Pain scores will be assessed using the 11-point VNRS (0 corresponding to no pain and 10 to the worst imaginable pain).

Transition from PACU to surgical ward will be considered to be safe when patient will achieved a Modified Aldrete Score ≥ 9. Although laparoscopic cholecystectomy is established as a day-case procedure, our protocol is designed to admit all patients for 24 h to ensure adequate follow-up of patients and for proper data collection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I-II patients
* 20-60 years

Exclusion Criteria:

* American Society of Anesthesiologists III and above patients
* BMI: 35 and above
* Hepatic, renal or cardiac insufficiency
* 2 degree Heart block and above
* Diabetes
* Psychiatric disease
* History of chronic pain
* Alcohol or drug abuse
* Allergy to any of a drug in the study groups
* Pregnant, breast-feeding or menstruating women
* Inability to use a patient-controlled analgesia device
* Any analgesic or antiemetic use in last 24 hours before anesthesia induction
* Any surgical complication that may affect the outcomes of the study (open surgery etc.)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Postoperative fentanyl consumption | 6 hours after extubation
  Patients will use a Patient controlled analgesia (PCA) device for 6 hours after extubation

SECONDARY OUTCOMES:
Recovery time | 2 hours after cessation of anesthesia infusions
  Extubation time after cessation of anesthesia infusions and discharge time from postanesthesia care unit (PACU) after extubation
Postoperative nausea and vomiting | Postoperative 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Faculty of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031